CLINICAL TRIAL: NCT03324295
Title: Aqueous Urea Concentration May be Related to Cataract Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hassan Lotfy Fahmy, Clinical Professor, Assiut University
Other Study IDs: IRB000078
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2017-10

CONDITIONS: Cataract Cortical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cortical cataract: patients with age related cortical cataracts who are otherwise healthy
  Interventions: Diagnostic Test: cortical cataract
- ocular problems: systemically healthy subjects with ocular problems other than cataract
  Interventions: Diagnostic Test: cortical cataract
- impaired renal functions: patients with impaired renal functions and are not on dialysis
  Interventions: Diagnostic Test: cortical cataract

INTERVENTIONS:
Diagnostic Test: cortical cataract — Blood urea

SUMMARY:
cataracts could be cured with eye drops. Some studies reported that in chronic renal failure, the occurrence of cataract is rare and the mechanism is unknown. The aim of this research is to describe correlation between urea concentration in the serum and aqueous humor and development of age related cataract.

DETAILED DESCRIPTION:
The study was conducted in the departments of Ophthalmology and internal medicine,

Asyut University hospitals, Egypt. Three groups of subjects were included:

patients with age related cortical cataracts who are otherwise healthy (cases) and two control groups; first systemically healthy subjects with ocular problems other than cataract and a second control group of patients with impaired renal functions and are not on dialysis treatment and thus have elevated serum urea levels. Slit lamp examination was performed to evaluate crystalline lens for opacities. Measurement of serum urea was done for all study subjects. Aqueous humor urea concentration was done only for the group of patients who are planned to have intraocular surgery. For that purpose, 0.1 ml of aqueous humor will be aspirated at the start of routine intraocular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Senile Cortical cataract.

Exclusion Criteria:

* Senile Nuclear cataract.
* Congenital cataract
* Traumatic cataract

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Assiut university hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Blood urea level | 1 Day
  The relation between blood urea level and cataract

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Fahmy, prof, Principal Investigator — Assiut University
Locations (1):
- Hassan Lotfy, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided